CLINICAL TRIAL: NCT02110277
Title: Photoacoustic Imaging of the Ovary
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr Zhu, collaborator and the inventor of the photoacoustic system, is leaving the institution and it is not feasible to conduct the study without the machine.
Sponsor: UConn Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Molly Brewer, Professor, Obstetrics and Gynecology, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-139S-3; R01CA151570 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2017-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Epithelial ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAI/ultrasound Diagnostic Group (Experimental): These patients will include women who are at risk for ovarian cancer and wish to undergo prophylactic oophorectomy, or who have an ovarian mass suggestive of a malignancy and are counseled to undergo oophorectomy.
  Interventions: Device: PAI/ultrasound Diagnostic Group

INTERVENTIONS:
Device: PAI/ultrasound Diagnostic Group — These patients will include women who are at risk for ovarian cancer and wish to undergo prophylactic oophorectomy, or who have an ovarian mass suggestive of a malignancy and are counseled to undergo oophorectomy.

SUMMARY:
The purpose of this study is to develop technology to image the ovaries in order to better evaluate ovarian disease and to study how these experimental imaging techniques might work together or separately to improve our ability to detect ovarian cancer.

DETAILED DESCRIPTION:
Epithelial ovarian cancer causes the highest mortality of any of the gynecologic cancers although it is the second most common gynecologic malignancy. Ovarian cancer is not usually detected earlier than Stage III or IV because it is usually asymptomatic; yet survival is high with early stage disease. In addition, women with a pelvic mass noted on ultrasound that undergo oophorectomy have only a 1-3% risk of malignancy and thus 97-99% will be overtreated because of our inability to reliably differentiate benign from malignant masses with ultrasound. BRCA1 testing and family history will identify certain high-risk individuals who have a higher risk of malignancy and need a modality that will be more reliable in detecting early cancers to provide more accurate surveillance.We are developing a new transvaginal imaging device optimized for ovarian cancer detection, diagnosis and validated from ex vivo and in vivo clinical studies. This automated system may provide an early diagnostic tool for ovarian cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* All patients, twenty one years or older, referred to the University of Connecticut for conditions necessitating oophorectomy.
* Patients cannot be pregnant or wish to become pregnant.
* Willingness to participate in the study.

Exclusion Criteria:

* All Subjects who fail to meet the inclusion criteria are ineligible for the study.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Brewer, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PAI/Ultrasound Diagnostic Group
Started (Two participants enrolled and started but did not complete due to study premature termination.) | 2
Completed (no results obtained. study terminated prematurely.) | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated and no results were analyzed.
Arm/Group | PAI/Ultrasound Diagnostic Group
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: To Measure Photoacoustic Imaging (PAI)/Ultrasound Signature From Ovaries Prior to Surgery Using the Ratio of Deoxy/Oxy Hb
Description: To develop a method of analyzing PAI ovarian tissue images measuring oxy and deoxy hemoglobin as well as the ratio of deoxy/oxy Hb to recognize the presence of ovarian abnormalities and compare changes seen with ultrasound to changes seen with PAI.
Time Frame: 5 years
Population: Study prematurely terminated and no results analyzed.
Arm/Group | PAI/Ultrasound Diagnostic Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Pathologic Diagnosis and in Vivo Imaging
Description: To characterize the tissue images with pathologic diagnosis and to refine the system based on the characteristic features of in vivo imaging.
Time Frame: 5 years
Population: 0 participants analyzed since study was terminated prematurely.
Arm/Group | PAI/Ultrasound Diagnostic Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | PAI/Ultrasound Diagnostic Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No